CLINICAL TRIAL: NCT03297528
Title: Multiple Consolidation Chemotherapy and DLI Prevent Second Relapse in Patients With Relapsed Acute Leukemia After Allotransplant and Achieving Complete Remission After Induction Chemotherapy and DLI
Brief Title: Chemotherapy and DLI for Prevention of Second Relapse in Patients With Relapsed Acute Leukemia After Allotransplant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUPH2017-2-21
Record Dates: First submitted 2017-02-21; First posted 2017-09-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Donor Lymphocyte Infusion; Allogeneic Hematopoietic Stem Cell Transplantation; Acute Leukemia; Minimal Residual Disease; Graft-versus-host Disease; Relapse
MeSH Terms: conditions — Neoplasm, Residual; Graft vs Host Disease; Recurrence | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Participants receive chemotherapy and donor lymphocyte infusions based on the state GvHD, even the participants have a negative result of minimal residual disease (MRD). If the participants have no GvHD,they will receive chemotherapy and donor lymphocyte infusion until they develop GvHD.
  Interventions: Drug: donor lymphocyte infusion
- control group (No Intervention): Participants don't receive chemotherapy and donor lymphocyte infusion as long as they have a negative result of MRD,in dispite of whether or not GvHD.

INTERVENTIONS:
Drug: donor lymphocyte infusion — Participants in study group receive chemotherapy and donor lymphocyte infusion based on the state of GvHD, even they have a negative result of MRD. If participants in study group have no GvHD, they will receive chemotherapy and donor lymphocyte infusion until they develop GvHD. If the participants in study group have GvHD, they will be observed. But, the participants in control group don't receive chemotherapy and donor lymphocyte infusion as long as they have a negative result of MRD, in despite of whether or not GvHD.
  Other Names: chemotherapy
  Arms: study group

SUMMARY:
Patients with acute leukemia relapsing after allotransplant and who respond to anti-leukaemia interventions are at high-risk of a second relapse. Previous studies from investigators reported an association between a positive minimal residual disease (MRD)-test after transplant and an increased risk of subsequent relapse. Also, patients developing chronic graft-versus-host disease (GvHD) after receiving DLI (donor lymphocyte infusion)for leukemia relapse after a first allotransplant have a lower likelihood of a second relapse compared with similar patients not developing chronic GvHD. And, our previous study also reported patients with chronic GvHD after DLI was associated with a greater frequency of a negative MRD-test and lower likelihood of subsequent relapse compared with similar persons not developing chronic GvHD. Based on these data the investigators designed a randomized control study to determine whether giving additional consolidation chemotherapy and DLI might decrease likelihood of second relapse in persons without chronic GvHD or with a positive MRD-test after initial post-relapse therapy with induction chemotherapy and DLI.

ELIGIBILITY:
Inclusion Criteria:

* (1) acute leukemia in first complete or second complete remission;
* (2) relapse after an allotransplant;
* (3) had full or partial donor chimerism;
* (4) received re-induction chemotherapy and DLI and achieved a negative MRD-test.

Exclusion Criteria:

* (1) active GvHD
* (2) active infection
* (3) organ dysfunction

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a positive results of minimal residual disease that is evaluated by testing aberrant leukemia-associated immune phenotypes and WT1 mRNA levels. | one year
  Investigators use two strategies to test for minimal residual disease in bone marrow samples: (1) aberrant leukemia-associated immune phenotypes detected by 4 colour flow cytometry; and (2) WT1 mRNA levels detected by polymerase chain reaction.

SECONDARY OUTCOMES:
Number of participants who relapsed | one year
  Relapse was defined as recurrence of ≥5% bone marrow blasts or of ≥1 extra-medullary sites of leukaemia.
Number of surviving participants | one year
  The outcomes of participants are recored until one year

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jun Huang, Study Director — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology,Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided